CLINICAL TRIAL: NCT05951270
Title: The Effects of Apple Polyphenol Supplementation on Glucose Homeostasis in Prediabetic Individuals
Brief Title: Glucose Homeostasis and Apple Polyphenols
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting participants with prediabetes
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL77812.068.21
Record Dates: First submitted 2023-06-27; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: PreDiabetes; Impaired Glucose Tolerance; Glucose Metabolism Disorders
Keywords: Apple Polyphenols; Prediabetes; Glucose homeostase
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: The study conforms to a randomized, double-blinded, placebo-controlled parallel study design.
Who Masked: Investigator
Masking Description: All samples and data will be coded so that no personal information about the participant can be inferred. Each subject will be assigned an individual code that will be visible on the biological samples. The code will include a participant number in chronological order and a test day number in chronological order. In addition, the label of each sample will indicate the date of collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Twelve weeks of 1100 mg of apple polyphenol supplementation. At the start, middle and end of the study, several measurements will take place.
  Interventions: Dietary Supplement: Apple Polyphenols
- Control (Placebo Comparator): Twelve weeks of 1100 mg of maltodextrin. This product is an enzymatically converted potato starch. The flavor and color will have a similar/identical appearance and taste as all mentioned antioxidants.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Apple Polyphenols — ApplePhenon® is prepared from unripe green apples (malus domestica) and contains a large amounts of polyphenols. The supplement contains 63.8% procyanidins, 12.4% flavon-3-ols, 6.5% chalcones and 10.8% phenolcarboxylic acids
  Other Names: Applephenon
  Arms: Intervention
Other: Control — The placebo used in this study is 1100 mg maltodextrin (Avebe, Veendam, the Netherlands). This product is an enzymatically converted potato starch. The flavor and color will have a similar/identical appearance and taste as all mentioned antioxidants.
  Arms: Control

SUMMARY:
The primary objective is to investigate the effect of apple polyphenol supplementation for 12 weeks on glucose homeostasis in prediabetic individuals. Further, this study has three secondary objectives: 1) to investigate whether daily supplementation at breakfast and dinner with apple polyphenols for 12 weeks affects the rhythm of glucose uptake over the day and reduces fasting glucose levels and postprandial glucose peaks; 2) to determine the effect of daily supplementation with apple polyphenols for 12 weeks on biomarkers of metabolic health; 3) to assess whether daily supplementation with apple polyphenols for 12 weeks alters fecal SCFA concentrations and fecal microbiota composition.

DETAILED DESCRIPTION:
Study Design:

45 Prediabetic adults will be included in a double-blind randomized placebo-controlled trial. All volunteers will be subjected to a 12-week period during which an apple polyphenol supplement or placebo will be ingested at breakfast and dinner. An intervention period of 12 weeks with a third visit half way of the intervention has been chosen. After 6 weeks and at the end of the study microbiota composition is measured since dietary intervention of at least 6 weeks is required to be able to measure changes in microbial composition and metabolic health. The third visit will be scheduled to monitor protocol compliance and check the well-being of subjects. Concomitant medication will be recorded as well as adverse events. In addition, subjects will be reminded about the intake of the investigational product and difficulties to compliance will be discussed. Subjects will perform an oral glucose tolerance test, blood samples are taken and fecal samples will be collected at the start of the study, half-way and at the end of the intervention period. The oral glucose tolerance test will be performed to determine glucose tolerance. During the OGTT blood glucose samples will be collected at 30, 60, 90 and 120 minutes in order to determine area under the curve of glucose as primary endpoint for the glucose tolerance. The blood samples are taken to measure whole blood glucose, serum insulin, HbA1c, metabolic profile, antioxidant levels (protocol compliance) and SCFA. The fecal samples are collected to assess the fecal microbiota composition and fecal SCFA concentration. Finally, at the start of the intervention, and after the third visit an Abott FreeStyle Libre Pro Continuous Glucose Monitoring (CGM)(Hoofddorp, The Netherlands) sensor is inserted. The Abott FreeStyle Libre Pro CGM sensor will be injected and worn for a period of 14 days after which the subjects will visit for collecting the data for continuous glucose monitoring with a recorder. The Abott FreeStyle Libre Pro is intended for use with type 2 diabetic individuals but a recent study has validated its use in prediabetic individuals (50).The baseline continuous glucose monitoring needs to be completed before the intervention will be started.

Screening and pre-testing:

Prior to the study, volunteers' suitability to participate will be assessed in a single screening session. The participants will be asked to come to the laboratory in fasted state (i.e. no eating or drinking after 22:00h the night before; drinking water is allowed) After explaining all study procedures, written informed consent will be obtained from subjects willing to participate. A signed copy of the informed consent will be provided for the subject to keep. The subject's suitability for the trial will be confirmed by the inclusion/exclusion criteria (see section 4). During screening, body weight, height and BMI (using the equation BMI = body mass (kg)/height (m)2 ) will be assessed. Subjects will be asked to fill in a medical questionnaire enquiring about their general health, medical history, GI symptoms, use of medication and sports activities. HbA1C will be measured using an Abbott™ Afinion™ 2 Analyzer (Hoofddorp, The Netherlands). Subjects will be included based on the results from BMI, and the in- and exclusion criteria discussed in the medical questionnaire. Included subjects will be instructed to collect a fecal sample to determine microbial composition- and activity and SCFA concentration. A collection kit will be provided to take home that includes a toilet hat, instructions for collecting the specimen, a collection tube, and a biohazard mailing bag. A short questionnaire about the collection time and date will be included in the collection kit as well as a dietary recall questionnaire. Food records and stool characteristics will be scored with a questionnaire and handed in by the subject at visit 1 (pre-test), as well as a fecal donation to determine microbial composition- and activity and SCFA concentration.

Test day:

Volunteers will visit the laboratory on six occasions over a twelve-week period. All subjects will be asked to record their dietary intake at three consecutive days in a food diary and to consume similar foods during the experimental period. Participants will be asked to record this in a food diary and approximately match caloric intake on the day prior to the second test day and eat the same type of meal. For the oral glucose tolerance test (OGTT), participants will be asked to come to the laboratory in fasted state (i.e. no eating or drinking after 22:00h the night before; drinking water is allowed), the participants will receive a standardized meal ("Aviko meal pan", Aviko bv. The Netherlands) from the researchers and the participants need to consume this meal prior to the OGTT testing days. The meals that the participants receive have a similar macronutrient composition and energy density. In addition, the food intake during the 3 days before the OGTT is asked to be kept similar. Participants need to abstain from strenuous exercise to maintain muscle glycogen stores and alcohol consumption for at least 48 h. Subjects perform the following experimental protocol three times, prior to, 39 to 45 and 81 to 87 days after the start of the intervention period. On arrival at the laboratory, subjects will be placed in a semi-supine position whilst a resting blood sample is collected from an antecubital vein (venipuncture) inserting a BC-shielded IV catheter. After providing the fasted blood sample, subjects will consume a glucose rich drink (75 grams corrected for weight). At 30-minutes, 60-minutes, 90-minutes and 120-minutes additional blood samples will be taken. An Abott FreeStyle Libre Pro will be injected for continuous glucose monitoring. The subjects will be asked to wear an Abott FreeStyle Libre Pro sensor for a period of 14 days. Subjects will be asked to collect the first three fecal samples after the OGTT. For this collection, participants will receive feces collection materials and collect the samples by themselves.

Intervention period:

Following the first OGTT, participants start the intervention period. During this 12-week intervention period, subjects will consume a supplement twice a day at breakfast and at dinner. Supplements contain either apple polyphenols (see section 5), or control, according to the randomization scheme. The intervention products are detailed in chapter 6. To facilitate participant compliance with adhering to the intake requirements and investigate the effect of antioxidants on the circadian pattern of glucose homeostasis, participants are advised to align their oral study product dosing to the timing of breakfast and dinner. In addition, a physical activity diary will be completed. At baseline and after 6 and 12 weeks of intervention, the following measurements will be performed: three-day food record, physical activity questionnaire, Bristol stool scores and Gastrointestinal Symptoms Rating Scores and a fecal sample. Subjects will be asked to maintain their regular exercise schema. Subjects will not receive individual results after measuring the outcome parameters, except when there will be unexpected findings (e.g. abnormal clinical parameter). Subjects can only participate in this study if they are willing to be informed about relevant unexpected findings (e.g. abnormal clinical parameter).

ELIGIBILITY:
Inclusion Criteria:

* Aged from 40 - 70 years
* 22.5 < BMI < 30 kg/m^2
* Weight-stable for at least 90 days prior to participation (no change in bodyweight, i.e. < 3kg).
* HbA1c: 5.7% to 6.4%
* Fasting blood glucose levels 100 to 125 mg/dl (5.6 to 6.9 mmol/l)

Exclusion Criteria:

* Subject following an overly imbalanced or restrictive diet as per nutritional advice
* Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be detrimental for the participants safety or potentially interfering with the study procedures and/or study outcome
* Abdominal surgery interfering with gastrointestinal function, upon judgement of the medical doctor, who will decide in-or exclusion based on the surgery applied
* Participants who received antibiotics in the 90 days prior to the start of the study
* Use of other medication will be reviewed by a medical doctor, who will decide on in- or exclusion based on the drug(s) used
* Use of laxatives within 14 days prior to the study
* Using medications for gastric or intestinal complaints
* Drug use, interfering with any of the outcome parameters of this study; to be decided by the person who is medically responsible for this study
* Having donated blood in the 3 months prior to the study
* Administration of antioxidant supplements, investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principle investigator), in the 14 days prior to the study
* History of side effects towards intake of antioxidant supplements
* Participants who have a gluten or lactose intolerance
* Use of proton pump inhibitors

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Apple polyphenols and glucose homeostasis in prediabetics | 12 weeks
  The primary outcome measure is the difference in glucose tolerance before and after the intervention, assessed using the oral glucose tolerance test area under the curve. Participants will undergo three oral glucose tolerance tests during the study: at the beginning, halfway, and the end. Prior to each test, participants will fast for at least 12 hours, consume a normal diet with approximately 150 grams of carbohydrate per day for three days, and avoid strenuous exercise and alcohol for at least 48 hours. During the test, participants will drink a glucose solution and have blood samples taken at various time points (0, 30, 60, 90, and 120 minutes) for analysis of glucose and insulin levels. Fasting insulin and glucose concentrations will be used to calculate insulin sensitivity using the homeostasis model assessment of insulin resistance (HOMA-IR) index. Blood samples will be stored for future use.

SECONDARY OUTCOMES:
Apple polyphenols and circadian pattern of blood glucose levels | 12 weeks
  For continuous glucose monitoring, for each participant, two times, at the beginning and end of the study a FreeStyle Libre Pro sensor will be applied. The investigator will insert the sensor in the participant using a sensor-applicator. The sensor will be inserted via a puncture and activated using a reader. The sensors will be worn for a period of 14 days after which the data are being collected by the investigator using the reader. The glucose concentrations over time will be obtained. Raw data will be analysed using an R-script. Using this script we can calculate the average blood glucose levels during the day and determine if the apple extract the observed glucose fluctuations over a 24 hour period.
Apple polyphenols and fecal microbiota composition | 12 weeks
  Measure the changes in microbiota composition after 12 weeks of apple extract supplementation. Participants will collect fecal samples at the beginning, halfway and at the end of the study.
  Fecal samples will be collected in dedicated feces collection tubes, which will be handed in by the subject to the investigator. Microbiota composition profiling will be done by HiSeq sequencing of the V4 and V5-V6 regions of the 16S rRNA gene.. In short, DNA isolated from feces will be used for amplification of the V4 and V5- V6 regions of the collective 16S rRNA genes using barcoded primers and fecal DNA as target. Afterwards, the NG-Tax pipeline will be used for microbiota profiling. Metabolite analysis will be done by organic acid HPLC. A variety of programs and in-house scripts will be used for bioinformatics analyses and multivariate statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Troost, Doctor, Principal Investigator — Maastricht University
Locations (1):
- Villa Flora, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
I will make the following end products available for further research and verification
  * Syntaxes
  * Documentation of the research process, including documentation of all participants
  * Data documentation (Several versions of) processed data
  * Raw data I will select a data format, which will allow other researchers and their computers (machine actionable) to read my data collection.
  Text documents --> PDF/A (.pdf) Spreadsheets --> CSV (.csv) Statistical data --> SPSS (.dat/.sps), R The data collection of my project will be findable for subsequent research. Data can be found through the search engine of the archive or repository in which it is stored. The data will be made findable for subsequent research. I will be using a persistent identifier as a permanent link to my data collection. Once the associated article is published and/or the project has ended, (part of) my data will be accessible for further research and verification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year end of study: before 03-02-2024.
Access Criteria: I have a set of terms of use available to me, which I will use to define the requirements of access to my data collection once the project has ended.
  * The permitted period of use of the data set
  * The manner in which the data set can be accessed
  * Person(s) who is/are authorised to give access to the data collection
  * The approval of the participants allows for further research using this data set
  * Conditions related to data security